CLINICAL TRIAL: NCT00678145
Title: Mechanisms of Hypoglycemia Associated Autonomic Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Meredith Hawkins, Principal Investigator, Albert Einstein College of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012-665; R01DK079974 (NIH)
Record Dates: First submitted 2008-05-14; First posted 2008-05-15 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus; Hypoglycemia; Autonomic Failure
Keywords: Diabetes; Hypoglycemia; HAAF; Counterregulation
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Pure Autonomic Failure | interventions — Naloxone; Fructose; Insulin; Exercise; Morphine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy (Experimental): Healthy individuals will receive drug (naloxone, morphine sulfate, epinephrine) and placebo comparator.
  Interventions: Drug: naloxone; Dietary Supplement: fructose; Behavioral: exercise; Drug: Morphine sulfate; Drug: Epinephrine
- Type 1 Diabetes (Experimental): T1D individuals will receive drug (naloxone, morphine sulfate, epinephrine) and placebo comparator.
  Interventions: Drug: naloxone; Dietary Supplement: fructose; Behavioral: exercise; Drug: Morphine sulfate; Drug: Epinephrine

INTERVENTIONS:
Drug: naloxone — Administering naloxone on Day 1, and quantifying the counterregulatory responses to hypoglycemia on Day 2.
  Other Names: Narcan
Dietary Supplement: fructose — Administering fructose on Day 1, and quantifying the counterregulatory responses to hypoglycemia on Day 2.
  Other Names: Insulin
Behavioral: exercise — Administering exercise on Day 1, and quantifying the counterregulatory responses to hypoglycemia on Day 2.
Drug: Morphine sulfate — Administering morphine on Day 1, and quantifying the counterregulatory responses to hypoglycemia on Day 2.
  Other Names: Morphine
Drug: Epinephrine — Administering epinephrine on Day 1, and quantifying the counterregulatory responses to hypoglycemia on Day 2.
  Other Names: Adrenalin

SUMMARY:
Intensive glucose control in type 1 diabetes mellitus (T1DM) is associated with clear health benefits (1). However, despite development of insulin analogs, pump/multi-dose treatment and continuous glucose monitoring, maintaining near-normal glycemia remains an elusive goal for most patients, in large part owing to the risk of hypoglycemia. T1DM patients are susceptible to hypoglycemia due to defective counterregulatory responses (CR) characterized by: 1) deficient glucagon release during impending/early hypoglycemia; 2) additional hypoglycemia-associated autonomic failure (HAAF) and exercise-associated autonomic failure (EAAF) that blunt the sympathoadrenal responses to hypoglycemia following repeated episodes of hypoglycemia or exercise as well as degrading other CR; and 3) hypoglycemia unawareness (HU), lowering the threshold for symptoms that trigger behavioral responses (e.g. eating). Thus, the risk of hypoglycemia in T1DM impedes ideal insulin treatment and leads to defaulting to suboptimal glycemic control (2). There are two approaches that could resolve this important clinical problem: 1) perfection of glucose sensing and insulin and glucagon delivery approaches (bioengineered or cell-based) that mimic normal islet function and precisely regulate glucose continuously, or 2) a drug to enhance or normalize the pattern of CR to hypoglycemia. Despite much research and important advances in the field, neither islet transplantation nor biosensor devices have emerged as viable long-term solutions for the majority of patients (3, 4). Over the past several years, our lab has explored the approach of enhancing CR by examining mechanisms responsible for HAAF/EAAF and searching for potential pharmacological methods to modulate the CR to hypoglycemia (5-11). Our work has led to a paradigm shift in the field of hypoglycemia, exemplified by the novel hypothesis and published experimental data supporting a role for opioid signaling that resulted in the initiation of exploratory clinical trials by other research groups.

DETAILED DESCRIPTION:
In the prior project period of R01 DK079974, we elucidated the central role played by the opioid signaling system as a mechanism for the development of HAAF/EAAF. We have demonstrated previously that opioid receptor blockade by acute infusion of naloxone during antecedent hypoglycemia can prevent experimentally induced HAAF in nondiabetic and T1DM subjects (JCEM 94:3372-80, 2009; JCEM 96:3424-31, 2011). We have also shown that opioid receptor blockade also abolishes EAAF, and that both effects are regulated by the stress response (hypoglycemia and exercise, respectively). Furthermore, recently we have shown that activation of μ-opioid receptors with IV infusion of morphine reproduces some of the key biochemical and clinical features of HAAF in nondiabetic humans.Taken together, these studies demonstrate that the opioid system plays a central role in hypoglycemia counterregulation and in HAAF.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic individuals

Exclusion Criteria:

* Hypertension
* Hyperlipidemia
* Heart disease
* Cerebrovascular disease
* Seizures
* Bleeding disorders

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2008-03 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Change in the counterregulatory responses to hypoglycemia compared to controls | Measured every 15 minutes at timepoints 0, 15, 30, 45...120 through study completion
  Measurements of counterregulatory hormones will be measured throughout the study

SECONDARY OUTCOMES:
Symptom scores | Measured every 15 minutes at timepoints 0, 15, 30, 45...120 through study completion
  Symptoms of hypoglycemia will be taken during the study

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Hawkins, M.D., M.S., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine / General Clinical Research Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carey M, Gospin R, Goyal A, Tomuta N, Sandu O, Mbanya A, Lontchi-Yimagou E, Hulkower R, Shamoon H, Gabriely I, Hawkins M. Opioid Receptor Activation Impairs Hypoglycemic Counterregulation in Humans. Diabetes. 2017 Nov;66(11):2764-2773. doi: 10.2337/db16-1478. Epub 2017 Aug 31. PMID 28860128
- [Derived] Milman S, Leu J, Shamoon H, Vele S, Gabriely I. Opioid receptor blockade prevents exercise-associated autonomic failure in humans. Diabetes. 2012 Jun;61(6):1609-15. doi: 10.2337/db11-1622. Epub 2012 Apr 20. PMID 22522612